CLINICAL TRIAL: NCT01254786
Title: Comparative Study of the Non-dependent Continuous Positive Pressure Ventilation and High Frequency Positive Pressure Ventilation During One-lung Ventilation for Thoracoscopy
Brief Title: Non-dependent HFPPV Versus CPAP for Video-assisted Thoracoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal University (Other)
Responsible Party: Dr. Mohamed El Tahan, University of Dammam
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201013
Record Dates: First submitted 2010-11-22; First posted 2010-12-07 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Elective Video-assisted Thoracoscopic Surgery; One-lung Ventilation Lasts at Least One Hour
Keywords: VATS; one lung ventilation; continuous positive pressure ventilation; high frequency positive pressure ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP2 - HFPPV group (Active Comparator): the non-dependent lung will be ventilated with CPAP of 2 cm H2O for 30 min followed with HFPPV for min.
  Interventions: Procedure: Non-dependent lung ventilation
- HFPPV-CPAP2 group (Active Comparator): the non-dependent lung will be ventilated with HFPPV for 30 min followed with CPAP of 2 cm H2O for 30 min.
  Interventions: Procedure: Non-dependent lung ventilation

INTERVENTIONS:
Procedure: Non-dependent lung ventilation — the dependent lung will be ventilated with conventional ventilation (OLV) a tidal volume of 6 mL/kg (predicted body weight), whereas FiO2, I: E ratio, PEEP, frequency, peak inspiratory pressures, and a flow of fresh gas will be maintained as during two-lung ventilation for 15 min.
  Then the non-dependent lung will be allowed to deflate to a CPAP of 2 cm H2O, which will be connected to the flowmeter of an oxygen cylinder with a flow rate of 5 L/min and FiO2 of 1.0 for 30 min
  Then, the non-dependent lung will be connected to a second identical ventilator, 15 min after OLV, using a FiO2 of 1.0, VT 3 mL/kg (predicted body weight), I: E ratio <0.3 and R.R 60 breaths/min for further 30 min.
  Arms: CPAP2 - HFPPV group
Procedure: Non-dependent lung ventilation — the dependent lung will be ventilated with conventional ventilation (OLV) a tidal volume of 6 mL/kg (predicted body weight), whereas FiO2, I: E ratio, PEEP, frequency, peak inspiratory pressures, and a flow of fresh gas will be maintained as during two-lung ventilation for 15 min.
  Then, the non-dependent lung will be connected to a second identical ventilator, 15 min after OLV, using a FiO2 of 1.0, VT 3 mL/kg (predicted body weight), I: E ratio <0.3 and R.R 60 breaths/min for further 30 min.
  Then the non-dependent lung will be allowed to deflate to a CPAP of 2 cm H2O, which will be connected to the flowmeter of an oxygen cylinder with a flow rate of 5 L/min and FiO2 of 1.0 for 30 min
  Arms: HFPPV-CPAP2 group

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) is usually performed using well-collapsed lung is essential for optimum surgical visualization and resection. However, one lung ventilation (OLV) is associated with deleterious impaired oxygenation secondary to the increases in shunt fraction.1 There are different approaches for the recruitment of the non-dependent lung (NL) during OLV such as the selective application of continuous positive pressure ventilation (CPAP) or high frequency positive pressure ventilation (HFPPV) to the non-dependent lung.2-4 These strategies may improve arterial oxygenation and reduce shunt fraction,2-4 However, the use of high CPAP levels impaired the surgical conditions during thoracotomy.2-3 On contrary, the application of HFPPV either to both lungs5or to the non-dependent lung permits adequate surgical conditions during thoracotomy.4 The investigators hypothesize that the application of volume-controlled HFPPV to the non-dependent lung during OLV for video-assisted thoracoscopic surgery may provide better surgical field and adequate oxygenation than the use of CPAP 2 cm H2O.

The investigators will evaluate the effects of the selective application of conventional one lung ventilation, HFPPV, or CPAP 2 cm H2O to the non-dependent lung on surgical field conditions, and arterial oxygen and carbon dioxide tensions (PaO2 and PaCO2, respectively) during OLV in the patients scheduled for video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Thirty patients aged 18-60 years (ASA physical status II-III) scheduled for elective video-assisted thoracoscopic surgery with at least one hour of one-lung ventilation (OLV) will be included in this randomized prospective placebo-controlled crossover study at the authors' center after obtaining approval of the institutional ethical committee and informed written consent. The patients will be randomized to a CPCP2-HFPPV group(n = 15)or a HFPPV-CPAP2 group(n = 15).

A power analysis of the data obtained from our preliminary pilot study indicated that 26 patients will be sufficient to detect a one SD changes in the visual analog scale assessment of the surgical field, with a type-I error of 0.05 and a power of 85%, with added 10% more patients, for a final sample size of 30 patients to account for patients dropping out during the study. All operations will be performed by the same surgeons.

The patients will be premedicated with fentanyl (1.0 μg/Kg) and i.v. midazolam (0.03 mg/Kg). All patients will be monitored with five leads electrocardiography, pulse oximetry, and non-invasive blood pressure and 7mL/Kg of 6% Hydroxyethyl Starch 130/0.4 (Voluven, Fresenius Kabi, Bad Homburg, Germany) will be given intravenously before induction of general anesthesia. An arterial line (20 G) will be inserted under local anesthesia. A thoracic epidural catheter (T4-T7) will be inserted with the patient in sitting position, and a test dose (1.5% lidocaine 3 mL plus epinephrine 1:200.000) will be administered in order to exclude an intravascular or intrathecal position of the catheter. No more epidural local anesthetics will be used during the study in order to avoid effects on hypoxic pulmonary vasoconstriction.

Anesthesiologists who gave the anesthetic will not be involved in the collection of the patient's data. General anesthesia will be induced with propofol (2-3 mg/kg), fentanyl (2-3 µg/kg), and cisatracurium (0.2 mg/kg) was given for muscle relaxation.

The trachea will be intubated with a left-sided double-lumen tube (DLT) [Broncho-Cath®; Mallinckrodt Medical Ltd., Dublin, Ireland]. The correct position of the tube will be confirmed with a fiberoptic bronchoscope after intubation and after positioning the patient in the lateral decubitus position. Other patient monitoring included end-tidal CO2, neuromuscular blockade, and nasopharyngeal temperature will be used. Anesthesia will be maintained with continuous infusions of propofol (6-8 mg/kg/h) and fentanyl (1 µg/kg/h). Increments of cisatracurium (0.03 mg/kg) will be given to maintain suppression of the second twitch using a train-of-four stimulation.

In all patients,the patients' two lungs will be mechanically ventilated with intermittent positive pressure ventilation using fraction of inspired oxygen (FiO2) of 0.5 in air, tidal volume (VT) of 8 mL/kg (predicted body weight), inspiratory to expiratory [I: E] ratio of 1:2.5, a positive end-expiratory pressure (PEEP) of 5 cm H2O, respiratory rate (R.R) will be adjusted to achieve an arterial carbon dioxide tension (PaCO2) 35-45 mm Hg, peak inspiratory pressures will be limited to 35 cm H2O and a low flow of fresh gas (<2 L/min) in a semi closed circuit system.

After positioning of the patient in the lateral decubitus position,the dependent non-operative lung will be ventilated conventionally(OLV)with a tidal volume of 6 mL/kg (predicted body weight), whereas FiO2, I: E ratio, PEEP, frequency, peak inspiratory pressures, and a flow of fresh gas will be maintained as during two-lung ventilation and the lumen of the non-dependent operative lung will be left open to air.

The subjects will be allocated randomly to two groups (n=15 each) by drawing sequentially numbered sealed opaque envelopes containing a computer-generated randomization code.

In CPAP2-HFPPV group, the non-dependent lung will be allowed to deflate to a CPAP of 2 cm H2O for 30 min, using a CPAP circuit (Bronchocath® CPAP system; Mallinckrodt Medical, Inc., St. Louis, MO) which will be connected to the flowmeter of an oxygen cylinder with a flow rate of 5 L/min and FiO2 of 1.0.7 Then, the lumen of non-dependent lung will be connected to a second identical ventilator with low compliant internal circuit. HFPPV will be initiated for 30 min using a FiO2 of 1.0, VT 3 mL/kg (predicted body weight), I: E ratio <0.3 and R.R 60 breaths/min.

In HFPPV-CPAP2 group, the non-dependent lung will be ventilated using HFPPV of the non-dependent lung for 30 min followed with non-dependent lung CPAP of 2 cm H2O for 30 min,

At the end of surgery, the nondependent lung will be re-expanded and two-lung ventilation will be resumed with a tidal volume of 8 mL/kg (predicted body weight). Twenty minutes before the skin closure, the infusions of propofol and fentanyl will be gradually decreased by 20% in every 5 minutes. At the end of surgery, the infusions will be discontinued, the residual neuromuscular block will be antagonized with neostigmine 50 μg/kg and atropine 20 μg/kg, and the patient will be extubated by the same anesthesiologists.

The surgical field conditions, oxygenation and hemodynamic data will be recorded after induction of general anesthesia (baseline), 15 (NL-15), 30 (NL-30) and 60 minutes (NL-60) after the selective application of CPAP or HFPV to the nondependent lung, and 15 min after returning of two-lung ventilation (TLV).

The surgeons will be asked to rate their satisfaction with the surgical field using a 10-cm VAS (0: worse; 10: excellent field). The ICU and hospital lengths-of-stay will be recorded.

Perioperative hypoxemia (SaO2<90%), respiratory and cardiovascular events, and mortality will be recorded within 30 days of surgery because a shorter period may have missed complications and deaths directly related to events that occurred after thoracic surgery.

Statistical analysis will be performed using the Statistical Package for the Social Sciences (Release 16, SPSS Inc., Chicago, IL, 2007). Data will be tested for normality using the Kolmogorov-Smirnov test. Repeated-measures analysis of variance will be used for analysis of serial changes in the patients' data at different times after the start of study intervention. Chi-square test will be used for categorical data. Dependent t-test and ANOVA will be used for continuous parametric variables. The Mann-Whitney U test will be performed for intergroup comparisons for the non-parametric values. Data will be expressed as mean (SD), number (%), or median [range]. A value of P<0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* elective video-assisted thoracoscopic surgery with at least one hour of one-lung ventilation (OLV)

Exclusion Criteria:

* decompensated cardiac diseases(>New York Heart Association II)
* pulmonary diseases(vital capacity or FEV1% < 50% of the predicted values)
* hepatic diseases
* renal diseases
* arrhythmias
* pulmonary hypertension (mean pulmonary artery pressure >30 mm Hg)
* previous history of pneumonectomy
* bilobectomy
* lobectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale rating of the surgical field conditions | every 15 min from the start of surgery
  Visual analog Scoring assesment of the surgical field conditions will be rated by the surgeons. VAS of 10 denotes the best surgical fied and VAS of 0 attributes inability to proceed with surgery

SECONDARY OUTCOMES:
Hemodynamic variables | every 15 min from the start of surgery
  hemodynamic parameters (heart rate and mean arterial blood pressure)
Respiratory variables | every 15 min from the start of surgery
  Respiration parameters (arterial carbon dioxide tensions (PaCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, M.D., Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- King Fahd hospital of the University of Dammam, Khobar, Eastern Province, Saudi Arabia